CLINICAL TRIAL: NCT03301389
Title: Cardiac Magnetic Resonance for Early Detection of Chemotherapy or Radiation Therapy Induced Cardiotoxicity in Breast Cancer (CareBest)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0730
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Chemotherapy Induced Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control group
  Interventions: Other: Cardiac magnetic resonance imaging
- Pretreatment group: Patients in pretreatment state
  Interventions: Other: Cardiac magnetic resonance imaging
- Anthracycline-based chemotherapy (3 months): Patients who received anthracycline-based chemotherapy 3 months ago
  Interventions: Other: Cardiac magnetic resonance imaging
- Anthracycline-based chemotherapy (6 months): Patients who received anthracycline-based chemotherapy 6 months ago
  Interventions: Other: Cardiac magnetic resonance imaging
- Anthracycline-based chemotherapy (more than 1 year ago): Patients who received anthracycline-based chemotherapy more than 1 year ago
  Interventions: Other: Cardiac magnetic resonance imaging
- Other therapy group: Patients who have been treated with other therapies (other chemo-therapies, combined radiation therapy, target agent therapy, hormone therapy)
  Interventions: Other: Cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Cardiac magnetic resonance imaging — The cardiac imaging protocol will include pre-contrast T1, post-contrast T1, and T2 mapping images acquired of the mid ventricle with the short axis plane for the analysis of native T1, T2, and extracellular volume (ECV) values of the myocardium. It will also include cine imaging covering the whole LV myocardium in the short axis plane for a functional analysis of the LV myocardium.

SUMMARY:
Chemotherapy or radiation therapy-induced cardiotoxicity are well-recognized side effects in patients with cancer. The clinical significance of cardiotoxicity is growing with increasing cancer survivor-ship.

Left ventricular (LV) functional assessment is the standard of reference to diagnose chemotherapy- or radiation therapy-induced cardiotoxicity. The investigators will investigate the usefulness of T1 mapping parameters for early detection and prediction of chemotherapy-, radiation therapy-, or other therapy-induced cardiotoxicity in breast cancer patients This study aimed to achieve early detection of chemotherapy- or radiation therapy-induced cardiotoxicity using T1 mapping magnetic resonance imaging (MRI) and determine a prognostic imaging factor of chemotherapy- or radiation therapy-induced cardiotoxicity in patients treated for breast cancer.

DETAILED DESCRIPTION:
Screening and follow-up cardiac magnetic resonance imaging (CMR) protocols for diagnosis of cardiotoxicity will be conducted in patients with breast cancer who have received or are planned to receive treatment for breast cancer. The protocol will include T1 and T2 mapping and cine imaging of the LV myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast cancer

Exclusion Criteria:

* Contraindication of MRI
* Failure with informed consent
* Fail to scan screening protocol

Ages: 17 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The breast cancer patient with pretreatment state The breast cancer patients with the prior chemotherapy, or radiation therapy The breast cancer patients receiving prior chemotherapy, or radiation therapy The breast cancer patients with other treatments
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in LVEF (left ventricular ejection fraction) | 1 year after CMR scanning
  Decrease in LVEF : more than 10% compared to the baseline LVEF) or LVEF < 50%
Decrease in LVEF (left ventricular ejection fraction) | 2 years after CMR scanning
  Decrease in LVEF : more than 10% compared to the baseline LVEF) or LVEF < 50%

SECONDARY OUTCOMES:
MACE (Major adverse cardiac events) | 1 year after CMR scanning
MACE (Major adverse cardiac events) | 2 years after CMR scanning

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Research Institute of Radiological Science, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong YJ, Han K, Lee HJ, Hur J, Kim YJ, Kim MJ, Choi BW. Assessment of Feasibility and Interscan Variability of Short-time Cardiac MRI for Cardiotoxicity Evaluation in Breast Cancer. Radiol Cardiothorac Imaging. 2024 Feb;6(1):e220229. doi: 10.1148/ryct.220229. PMID 38329404
- [Derived] Hong YJ, Kim GM, Han K, Kim PK, Lee SA, An E, Lee JY, Lee HJ, Hur J, Kim YJ, Kim MJ, Choi BW. Cardiotoxicity evaluation using magnetic resonance imaging in breast Cancer patients (CareBest): study protocol for a prospective trial. BMC Cardiovasc Disord. 2020 Jun 3;20(1):264. doi: 10.1186/s12872-020-01497-y. PMID 32493217